CLINICAL TRIAL: NCT01422070
Title: A Multi-centre European Observational Study to Assess Whether Patients Admitted to the ICUs With Availability of Intermediate Care Unit (IMCU) Have Lower Hospital Mortality Than Those Admitted to the ICUs Without Availability of IMCU
Brief Title: European Mortality & Length Of Intensive Care Unit (ICU) Stay Evaluation (ELOISE)
Acronym: ELOISE
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: University Hospital of Ferrara (Other); European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Maurizia Capuzzo, Medical Doctor, Università degli Studi di Ferrara
Other Study IDs: 80-2011
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-07

CONDITIONS: Critical Illness
Keywords: mortality; intensive care; critical care; intermediate care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients admitted to the Study Units: Consecutive adult patients consecutively admitted to the Study Units during one month (either from 7th November to 4th December 2010, or from 16th January to 12th February 2012)

SUMMARY:
The starting point of ELOISE is the significant number of Intensive Care Unit (ICU) survivors who die after the transfer to ward. This mortality rate nullifies the sophisticated diagnostics and the life-support therapies adopted in the ICU.

The inadequate care available at the destination ward has been suggested as one of the reasons to explain the bad outcome of some ICU survivors, but most hospitals do not have enough ICU beds to prolong the ICU stay until the patient has fully recovered. Therefore, Inter Mediate Care Units (IMCU) with levels of nursing staff and costs lower than ICU but higher than wards have been proposed to facilitate discharges of ICU patients. Unfortunately the literature does provide evidence of efficacy of IMCU.

The primary aim of the study is to assess whether the patients admitted to ICUs with availability of IMCU have lower hospital mortality than those admitted to the ICU without availability of IMCU.

Secondary aims are as follows:

1. To compare Lengths Of ICU and Hospital Stay (LOIS and LOHS, respectively) of patients admitted to ICUs with or without availability of IMCU.
2. To assess the influence of IMCU on the rate of ICU readmissions.
3. To compare the hospital survival of patients discharged to IMCU and general ward (in hospital with or without availability of IMCU) adjusted for severity of illness and nursing workload at ICU discharge. This last aim will require a larger sample size (more than 10,000), but we hope to collect such a sample.

DETAILED DESCRIPTION:
Despite the high cost of Intensive Care Unit (ICU), a significant number of patients surviving intensive care die subsequently in hospital after the transfer to ward. Mortality rates after discharge from ICU have been reported to range from 6.1 to 27%

In 2000, it was reported that premature discharge from ICU was more likely to occur at night and was associated with higher death rates. Suggested factors that might account for a worse outcome for night discharges were poorer quantity and quality of care available at night both during transfer and at the destination. The implication of this study for the health system was that many hospitals did not have enough ICU beds. To facilitate earlier ICU discharges of ICU patients who are thought to need more care than those which can be provided on wards, InterMediate Care Units (IMCU) with level of nursing staff (and costs) lower than ICU were proposed more than a decade ago.

Despite the relevance of the topic, the literature on the efficacy and cost-effectiveness of IMCU available at present shows variable results. And the potential benefits of IMCUs remain uncertain.

The most striking are probably the following questions:

* Does IMCU decrease the hospital mortality rate of ICU patients?
* Does IMCU allow earlier ICU discharge and hence improve patients flux through the ICU and reduce ICU cost?
* Does IMCU permit a reduction of ICU readmissions? We propose to address these issues in a large multinational, multicentre study.

ELIGIBILITY:
Inclusion Criteria:

* admission to one of the Study Unit
* any organ support allowed
* age of at least 16 years

Exclusion Criteria:

* age lower than 16 years
* patients admitted as donor for transplant
* patients admitted with limitation of care stated before admission

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients consecutively admitted to the Study Units during one month (from 7th November to 4th December 2010)
Sampling Method: Probability Sample
Enrollment: 6433 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizia Capuzzo, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Ferrara, Italy; Christophe Combescure, Statistician, Study Chair — University of Geneva, Switzerland; Bertrand Guidet, PhD, Study Chair — Hôpital Saint-Antoine, Paris, France; Gaetano Iapichino, MD, Study Chair — Hospital San Paolo, University of Milan, Italy; Paolo Merlani, MD, Study Chair — University of Geneva, Switzerland; Rui P Moreno, PhD, Study Chair — Hospital de Santo Antonio dos Capuchos, Lisbon, Portugal; Thomas Perneger, Statistician, Study Chair — University of Geneva, Switzerland; Andrew Rhodes, PhD, Study Chair — St George's Hospital, London, UK; Andreas Valentin, MD, Study Chair — University of Vienna, Austria
Locations (1):
- Maurizia Capuzzo, Ferrara, Italy

REFERENCES:
- [Result] Capuzzo M, Volta C, Tassinati T, Moreno R, Valentin A, Guidet B, Iapichino G, Martin C, Perneger T, Combescure C, Poncet A, Rhodes A; Working Group on Health Economics of the European Society of Intensive Care Medicine. Hospital mortality of adults admitted to Intensive Care Units in hospitals with and without Intermediate Care Units: a multicentre European cohort study. Crit Care. 2014 Oct 9;18(5):551. doi: 10.1186/s13054-014-0551-8. PMID 25664865
- [Derived] Poncet A, Perneger TV, Merlani P, Capuzzo M, Combescure C. Determinants of the calibration of SAPS II and SAPS 3 mortality scores in intensive care: a European multicenter study. Crit Care. 2017 Apr 4;21(1):85. doi: 10.1186/s13054-017-1673-6. PMID 28376908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All admissions of patients aged ≥ 16 years to a study during 28-day period (from 7 Nov to 4 Dec 2011, or from 16 Jan to 12 Feb 2012), excludind admissions only for organ donation, and with any limitation of care stated before unit admission. Maximum number of admissions per unit was 100.
Pre-assignment Details: Prospective observational study, without group assignment. Study units gave information about organization. 32 admissions to units with level of care lower than intensive care unit (ICU), 337 readmissions, 83 admissions out of the dates of enrollment slots, and 147 admissions with unknown vital status at hospital discharge were excluded.
Groups:
- Units in Hospitals With Intermediate Care Unit: Adult patients consecutively admitted to Intensive Care Units in hospitals with intermediate care unit
- Units in Hospitals Without Intermediate Care Unit: Adult patients consecutively admitted to Intensive Care Units in hospitals without intermediate care unit
Period: Overall Study
Arm/Group | Units in Hospitals With Intermediate Care Unit | Units in Hospitals Without Intermediate Care Unit
Started | 5031 (Number of patients admitted to 140 intensive care units) | 803 (Number of patients admitted to 27 intensive care units.)
Completed | 5031 | 803
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 337 readmissions, 83 admissions with inconsistencies in dates and 147 patients with unknown vital status at hospital discharge (82 still in hospital at 90 days and 65 with missing vital status) were excluded from the analysis.
Groups:
- Units With Intermediate Care Unit: Patients admitted to intensive care unit with intermediate care unit in the hospital
- Units Without Intermediate Care Unit: Patients admitted to intensive care unit without intermediate care unit in the hospital
- Total: Total of all reporting groups
Arm/Group | Units With Intermediate Care Unit | Units Without Intermediate Care Unit | Total
Number analyzed (Participants) | 5031 | 803 | 5834
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [52 to 75] | 68 [55 to 77] | 65 [53 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2002 | 332 | 2334
  Male | 3029 | 471 | 3500

OUTCOME MEASURES:

1. Primary Outcome: Vital Status at Hospital Discharge
Description: Hospital mortality of the patients admitted to intensive care units with or without intermediate care unit in the hospital
Time Frame: Max 90 days after admission to the Study Unit
Measure: Number; unit: participants
Groups:
- Units in Hospitals With Intermediate Care Unit: Patients admitted to intensive care unit with intermediate care unit in the hospital
- Units in Hospitals Without Intermediate Care Unit: Patients admitted to intensive care unit without intermediate care unit in the hospital
Arm/Group | Units in Hospitals With Intermediate Care Unit | Units in Hospitals Without Intermediate Care Unit
Number analyzed (Participants) | 5031 | 803
participants | 1232 | 165

2. Secondary Outcome: Length of ICU Stay
Description: Number of days (calendar days -1) from admission to and discharge from the Study Unit
Time Frame: Max 90 days after admission to intensive care unit
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Units in Hospitals With Intermediate Care Unit | Units in Hospitals Without Intermediate Care Unit
Number analyzed (Participants) | 5031 | 803
days | 3.7 [1.9 to 7.7] | 2.8 [1.8 to 4.8]

3. Secondary Outcome: Length of Hospital Stay
Description: Number of days (calendar days -1) from admission to the Study Unit to discharge from the hospital
Time Frame: Max 90 days after admission to the Study Unit
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Units in Hospitals With Intermediate Care Unit | Units in Hospitals Without Intermediate Care Unit
Number analyzed (Participants) | 5031 | 803
days | 13.9 [7.6 to 25.0] | 11.0 [6.2 to 11.0]

4. Secondary Outcome: Number of ICU Readmissions
Description: Number of readmissions to intensive care unit during the same hospital course
Time Frame: Max 90 days after admission to the Study Unit
Measure: Number; unit: readmissions
Arm/Group | Units in Hospitals With Intermediate Care Unit | Units in Hospitals Without Intermediate Care Unit
Number analyzed (Participants) | 5031 | 803
readmissions | 292 | 40
Statistical Analysis 1: Comparison: Units in Hospitals With Intermediate Care Unit vs Units in Hospitals Without Intermediate Care Unit; The null hypothesis was that hospital mortality of patients admitted to intensive care units with intermediate care unit in the hospital is similar to that of the patients admitted to intensive care units without intermediate care unit in the hospital; Test type: Superiority or Other; p < 0.05, generalized estimating equation; Generalized estimating equation adjusts the confidence interval for the correlation of outcomes within-centre; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.45 to 0.88] — The fully adjusted multivariable logistic regression analysis showed an OR of 0.63 in favour of the presence of an intermediate care unit in the hospital

ADVERSE EVENTS:
Description: Adverse events were not collected.
Groups:
- Adverse Events Not Collected: Adverse events were not collected
Arm/Group | Adverse Events Not Collected
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No